CLINICAL TRIAL: NCT05678764
Title: Evaluation of a Conversational Information Collection Tool to Access Talk Therapy
Status: Completed | Type: Observational
Sponsor: Limbic Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: 112233
Record Dates: First submitted 2022-12-23; First posted 2023-01-10 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Mental Health Issue

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Conversational Information Collection Tool Referrals: These are patients who refer to talk therapy using the novel information collection tool.
  Interventions: Device: Conversational Information Collection Tool
- Other Referrals: These are patients who refer to talk therapy using other referral methods.

INTERVENTIONS:
Device: Conversational Information Collection Tool — Conversational Information Collection Tool that facilitates the self-referral to talk therapy.
  Groups: Conversational Information Collection Tool Referrals

SUMMARY:
This is an observational study evaluating a conversational information collection tool to access talk therapy.

The patient outcome data will be compared between people who refer to talk therapy via the conversational information collection tool and people who refer using other means.

ELIGIBILITY:
Inclusion Criteria:

* Participant meets minimum age requirements for the talk therapy service Participant's registered GP is within the talk therapy service's CCG catchment area

Exclusion Criteria:

* Participants who are in crisis (defined by requiring urgent care or being at an urgent risk of harm)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who refer to the talk therapy services that use the conversational information collection tool.
Sampling Method: Non-Probability Sample
Enrollment: 104874 (Actual)
Dates: Start 2023-06-29 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-10-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline depression score to after treatment | The definition of reliable and clinically significant improvement is based on a comparison of pre-treatment (at time of referral, on the day of consenting) and post-treatment (assessed at point of discharge, an average of 5 months) clinical score.
  The primary outcome will be defined as reliable and clinically significant improvement in clinical scores after treatment. Hereby, the investigators will test for changes in depression scores using Patient Health Questionnaire-9 (PHQ-9: posttreatment scores <10 and improved by ≥6 points). PHQ-9 includes 9 questions scored between 0 and 3, with higher scores indicating more severe depression.
Change from baseline anxiety score to after treatment | The definition of reliable and clinically significant improvement is based on a comparison of pre-treatment (at time of referral, on the day of consenting) and post-treatment (assessed at point of discharge, an average of 5 months) clinical score
  The primary outcome will be defined as reliable and clinically significant improvement in clinical scores after treatment. Hereby, we will test for changes in anxiety scores using Generalised Anxiety Disorder Assessment (GAD-7: posttreatment scores <8 and improved by ≥4 points).GAD-7 includes 7 questions scored between 0 and 3, with higher scores indicating more severe anxiety.
Clinical assessment times | This measure will be available after the clinical assessment (up to average of 1 month from consenting).
  Improved clinical efficiency will be indicated by reduced assessment times, measured by the average time per clinical assessment (in minutes).

SECONDARY OUTCOMES:
Waiting times | This measure will be available after the clinical assessment (up to average of 1 month from consenting).
  Patient waiting times for treatment will be measured as the time between the date of (self-referral) and the date of the clinical assessment.
Referral Dropout Rates | During Information Collection Tool interaction (day 1)
  Patient referral dropout will be measured as any individual who consented to participate in the study, but did not complete all requested clinical information during the referral process.
Assessment Dropout Rates | At time point of treatment termination using standard IAPT definitions (assessed up to 3 months)
  Clinical assessment dropout will be measured as any cancellation or "Did Not Attend" event for patients who successfully had a clinical assessment slot (eg. time and date) organised. The treatment cohort (Limbic Access with AI pathway) will be evaluated against a cohort of patients going through limbic Access' standard pathway across the same services and over the same time window as the study will be used for comparison.
Treatment Dropout Rates | At time point of treatment termination using standard IAPT definitions (assessed up to 3 months)
  Treatment dropout will be measured using a "dropout" label which is added to a patient's file in the service's patient management system by the treating clinician when a dropout event occurs. The treatment cohort (Limbic Access +AI pathway) will be evaluated against a cohort of patients going through limbic Access' standard pathway across the same services and over the same time window as the study will be used for comparison.

CONTACTS AND LOCATIONS:
Locations (3):
- United Kingdom (3):
  - Surrey and Borders Partnership NHS Foundation Trust, Leatherhead, Surrey
  - Essex Partnership University NHS Foundation Trust, Epping
  - Lincolnshire Partnership NHS Foundation Trust, Lincoln

IPD SHARING:
Plan to Share IPD: Undecided
Fully anonymised data might be shared as part of the publication process.